CLINICAL TRIAL: NCT07068659
Title: Effects of Circuit Aerobic Training and Circuit Resistance Training on Cardiorespiratory Fitness, Cardiovascular Response, and Peak Expiratory Flow Rate in Autistic Spectrum Disorder Children
Brief Title: Circuit Aerobic Training and Circuit Resistance Training in Autistic Spectrum Disorder Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Lizza- REC/RCR&AHS 24/0365
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Autism
Keywords: Autism spectrum disorder; Cardiorespiratory fitness; Peak expiratory flow rate; Circuit Training
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Circuit Aerobic Training
  Interventions: Other: Circuit Aerobic Training
- Group B (Active Comparator): Circuit Resistance Training
  Interventions: Other: Circuit Resistance Training

INTERVENTIONS:
Other: Circuit Aerobic Training — Participant will start with five-minute warm-up consisting of running at a heart rate under 100 beats per minute, followed by stretching for 20 sec. For the 30-minute aerobic portion of the exercise sessions, in weeks 1 - 2, participants will be required to complete two circuits of walking for 5 minutes, stepping up and down on a 30 cm step for 4 minutes, and walking backward and forward for 10 meters for 5 minutes. In weeks 3 - 4, participants will complete two circuits of walking for 4 1/2 minutes, stepping up and down on a 30 cm step for 4 minutes, and walking backward and forward for 10 meters for 5 minutes. In weeks 5 - 6, participants will complete two circuits of walking for 5 minutes, stepping up and down on a 30 cm step for 5 minutes, and walking backward and forward for 10 meters for 5 minutes. The rest interval between the circuits will be 5 minutes and between the sets between 30 seconds. The intensity of the aerobic exercises will be maintained at 9 - 15 on the rating of
  Arms: Group A
Other: Circuit Resistance Training — Participant will start with five-minute warm-up consisting of running at a heart rate under 100 beats per minute, followed by stretching for 20 sec. For the 30-minute resistance portion of the exercise sessions, in weeks 1 - 2, participants will be required to complete two circuits of hamstring curl with ankle weight on each leg for 5 minutes, leg raises with ankle weight on each leg for 4 minutes, and modified squats with weights for 5 minutes. In weeks 3 - 4, participants will complete two circuits of hamstring curl with ankle weight on each leg for 4 1/2 minutes, leg raises with ankle weight on each leg for 4 minutes, and modified squats with weights for 5 minutes. In weeks 5 - 6, participants will complete two circuits of hamstring curl with ankle weight on each leg for 5 minutes, leg raises with ankle weight on each leg for 5 minutes, and modified squats with weights for 5 minutes. The rest interval between the circuits will be 5 minutes and between the sets between 30 seconds. Ch
  Arms: Group B

SUMMARY:
Autism Spectrum Disorder (ASD) is a developmental condition that impacts a child's ability to communicate and interact socially, often accompanied by repetitive behaviors and unique patterns of activity. In addition to these core characteristics, children with ASD frequently exhibit lower levels of physical fitness and are at risk for a range of health concerns, including compromised cardiovascular health and reduced respiratory function. These physical limitations can contribute to broader health disparities and reduced quality of life. Regular physical activity is increasingly recognized as an important element in managing these challenges, offering benefits that extend beyond physical health to improve social skills, behavior, and overall well-being. However, understanding which types of physical activity can most effectively enhance cardiorespiratory fitness and respiratory performance in children with ASD remains a developing field. Examining the effects of structured exercise programs, such as circuit training, can provide valuable insights into optimizing fitness strategies that cater to the unique needs of children on the autism spectrum. The objective of study is to determine the effects of circuit aerobic training and circuit resistance training on cardiorespiratory fitness, cardiovascular responses, and peak expiratory flow rate in Autistic spectrum disorder children It is a randomized clinical trial. A consecutive sampling technique will be used to recruit the ASD children for the study. Then, they will be divided into two groups by simple random sampling through sealed opaque enveloped. Hand Grip Exercise will be given as baseline treatment. In group A patients will be given with circuit aerobic training while in group B patients will be given with circuit resistance training. The 6-minute walk test will be used to assess cardiorespiratory fitness (VO2 max), peak expiratory flow meter will be used to check peak expiratory flow rate (PEFR), and digital sphygmomanometer will be used to check cardiovascular response. Data will be entered and analyzed through SPSS version 21.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is defined as a lifelong neurodevelopmental disorder characterized by two key symptoms: persistent deficits in social communication/interaction and restricted, repetitive patterns of behavior and abnormal sensory responses. The severity of these symptoms varies extensively from one patient to another, leading to a multitude of clinical presentations. Onset of ASD can usually be observed during childhood, with signs detectable as early as 18 months of age. However, ASD remains extremely challenging to diagnose due to the diversity of clinical presentations and diagnosis requires both awareness from parents and caregivers to detect signs and an assessment from a multidisciplinary medical/paramedical team to confirm signs.

The World Health Organization (WHO) estimates the international prevalence of ASD at 0.76%; however, this only accounts for approximately 16% of the global child population. The Centers for Disease Control and Prevention (CDC) estimates about 1.68% of United States (US) children aged 8 years (or 1 in 59 children) are diagnosed with ASD. ASD occurs in all racial, ethnic, and socioeconomic groups, but its diagnosis is far from uniform across these groups. ASD is more common in males but in a recent meta-analysis, true male-to-female ratio is closer to 3:1 than the previously reported 4:1, though this study was not done using the DSM-5 criteria. Studies of children with sex chromosome aneuploidy describe a specific social functioning profile in males that suggests more vulnerability to autism.

Several studies have indicated different treatment techniques used to minimize the effects and the intensity of the symptoms, including antecedent-based treatments, consequence-based treatments, extinction-based treatments, and combinations of treatment strategies, psychopharmalogical-based treatment, and the use of physical exercise. Studies have been demonstrated that physical exercise ameliorates deficits in social interaction, reduces aggressive behaviors, and reduces stereotypical behavior in children, teenagers, and adults with ASD. Circuit aerobic training consists of a sequence of cardiovascular exercises performed with minimal rest periods between sets, aiming to keep the heart rate elevated and improve endurance. This type of training typically includes activities such as jumping jacks, running in place, and step-ups, arranged to target different muscle groups while maintaining a high level of aerobic intensity. Research indicates that circuit aerobic training effectively enhances cardiorespiratory fitness by stimulating sustained energy expenditure and cardiovascular adaptation. The continuous nature of the exercises promotes an increased oxygen uptake and endurance capacity, making it a valuable component of fitness programs for improving overall aerobic health. Circuit resistance training involves a series of strength-focused exercises performed in a structured sequence with limited rest intervals. This method integrates various resistance exercises targeting major muscle groups, such as squats, push-ups, and weightlifting activities, designed to build muscular strength and endurance while maintaining an elevated heart rate. The approach not only contributes to muscle development but also fosters improvements in cardiovascular health due to its dynamic and fast-paced nature. Studies show that circuit resistance training supports muscle hypertrophy, enhances power, and improves metabolic efficiency, offering comprehensive benefits for both strength and cardiovascular conditioning.

The study on the "Effects of Circuit Aerobic Training and Circuit Resistance Training on Cardiorespiratory Fitness, Cardiovascular Responses, and Peak Expiratory Flow Rate in Autistic Spectrum Disorder Patients" possesses substantial societal worth. People with ASD often have difficulties with motor skills, physical activity, and health-related fitness, which affects their general quality of life significantly. Effective strategies to enhance cardiorespiratory fitness, cardiovascular health, and respiratory function in people with ASD could be found by investigating customized physical training regimens. Improvements in social interaction, mental stability, and physical health may encourage increased independence and participation in community events. In order to promote a more accepting and helpful society, healthcare professionals, educators, and carers may be encouraged to implement evidence-based fitness programs that enhance the physical well-being of individuals with ASD while simultaneously encouraging their cognitive and emotional growth.

ELIGIBILITY:
Inclusion Criteria:

* Age 7-17
* Diagnosed Autistic (ASD) Children with 2 gold standard test Autism Diagnostic Observation Schedule (ADOS) and the Autism Diagnostic Interview-Revised .
* Vineland scale-II completed by parents that assessed three dimensions of adaptive daily behaviors (communication, daily living skills and socialization), and children with average score between 85-115 out of total score 20-160 will be selected

Exclusion Criteria:

* Contra-indication against physical exercise (e.g., cardiovascular disease or cardiac insufficiency that might alter heart rate (HR) response)
* Psychiatric disorders or comorbid medical (e.g., no epilepsy)
* Severe osteo-articular pathology
* Respiratory disorders (e.g., asthma)
* Medical treatment that may alter the metabolic response
* Cognitive disabilities (IQ < 70)

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Peak Expiratory Flow Rate | Baseline, Week 3, Week 6
Modified Six Minute Walk Test | Baseline, Week 3, Week 6
Systolic Blood Pressure | Baseline, Week 3, Week 6
Disatolic Blood Pressure | Baseline, Week 3, Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Danish Hassan, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Toscano CVA, Ferreira JP, Quinaud RT, Silva KMN, Carvalho HM, Gaspar JM. Exercise improves the social and behavioral skills of children and adolescent with autism spectrum disorders. Front Psychiatry. 2022 Dec 22;13:1027799. doi: 10.3389/fpsyt.2022.1027799. eCollection 2022. PMID 36620673
- [Background] Hodges H, Fealko C, Soares N. Autism spectrum disorder: definition, epidemiology, causes, and clinical evaluation. Transl Pediatr. 2020 Feb;9(Suppl 1):S55-S65. doi: 10.21037/tp.2019.09.09. PMID 32206584
- [Background] Bougeard C, Picarel-Blanchot F, Schmid R, Campbell R, Buitelaar J. Prevalence of Autism Spectrum Disorder and Co-morbidities in Children and Adolescents: A Systematic Literature Review. Front Psychiatry. 2021 Oct 27;12:744709. doi: 10.3389/fpsyt.2021.744709. eCollection 2021. PMID 34777048